CLINICAL TRIAL: NCT00678119
Title: A Phase II Study Testing the Safety and Activity of AGS-003 as an Immunotherapeutic in Subjects With Newly Diagnosed Advanced Stage Renal Cell Carcinoma in Combination With Sunitinib
Brief Title: Study Testing the Biologic Activity and Safety of a Immunotherapeutic in Patients With Newly Diagnosed Advanced Stage Kidney Cancer in Combination With a Marketed Renal Cell Carcinoma Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-003-006
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney cancer; Renal cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1: AGS-003+sunitinib (Experimental): Single arm study AGS-003 plus sunitinib
  Interventions: Biological: AGS-003; Drug: Sunitinib

INTERVENTIONS:
Biological: AGS-003 — Dendritic cell Immunotherapeutic
Drug: Sunitinib — An approved drug for the treatment of RCC
  Other Names: Sutent

SUMMARY:
Study to investigate an anticancer cellular immunotherapeutic, AGS-003, when used in combination with sunitinib in subjects with previously untreated advanced stage RCC.

DETAILED DESCRIPTION:
The purpose of this study is to investigate an anticancer immunotherapeutic, AGS-003, when used in combination with sunitinib (the treatment regimen) in a single-stage, Phase II design in subjects with previously untreated advanced stage RCC after nephrectomy/excisional biopsy/metastasectomy. AGS-003 is formulated using mature DCs co-electroporated with CD40L IVT RNA and autologous total tumor RNA

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects ≥18 years of age with newly diagnosed advanced stage RCC will be eligible for inclusion in this study if all of the following criteria apply:

1. Newly diagnosed advanced stage RCC.
2. Eligible for unilateral nephrectomy or partial nephrectomy; OR, Has lesion accessible for excisional biopsy/metastasectomy.
3. Measurable disease.
4. Candidate for sunitinib treatment as labeled.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Memorial Sloan Kettering Cancer Center (MSKCC) risk group 0 or 1.
7. No brain metastases detected by MRI.
8. Normal renal function in the contralateral kidney.
9. Able to abstain from taking prohibited prescription or prohibited non-prescription drugs.
10. Use of appropriate birth control methods for the duration of the study for women of childbearing potential and men with female partners of childbearing potential.
11. Clinically acceptable Screening results according to the following specific limits:

    * Adequate hematologic function.
    * Adequate renal and hepatic function.
    * Adequate coagulation function.
12. Normal serum calcium.
13. Ability to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
14. Voluntary informed consent given to participate in the study.

Exclusion Criteria:

Subjects will NOT be eligible for inclusion in this study if any of the following criteria apply:

1. Nephrectomy for RCC therapy is required.
2. Any serious medical condition or illness considered by the investigator to constitute an unwarranted high risk for investigational treatment.
3. Uncontrolled hypertension.
4. Type I diabetes mellitus (insulin therapy for Type II diabetes IS permitted).
5. Prior systemic therapy for advanced stage RCC.
6. Active autoimmune disease.
7. Prior history of malignancy other than RCC within the preceding 5 years, except for adequately treated cervical cancer or non-melanoma skin cancer.
8. Use of prohibited prescription or prohibited non-prescription drugs during 2 months prior to entry into the study.
9. Active, acute, or chronic clinically significant infections.
10. Use of another investigational drug or participation in any investigational drug study within the 28 days prior to the start of study enrollment.
11. Planned or elective anti-cancer surgical treatment other than nephrectomy/excisional biopsy/metastasectomy.
12. History of hypercalcemia, symptomatic hypercalcemia, or hypercalcemia requiring management.
13. Known hypersensitivity to dimethyl sulfoxide (DMSO).
14. Body weight less than 30 kg.
15. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Clinical antitumor activity will be assessed as an objective tumor response as defined by RECIST. Tumor response is documented using standard definitions of CR and must be confirmed no less than 4 weeks after the criteria for response are first met. | 24 weeks

SECONDARY OUTCOMES:
The monitoring of clinical activity, immune response and safety across multiple doses. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fred Miesowicz, Study Director — Argos Therapeutics
Locations (14):
- United States (12):
  - City of Hope, Duarte, California
  - UCLA, Los Angeles, California
  - The Urology Center of Colorado, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - The Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Carolina's Medical Center / Blumenthal Cancer Center, Charlotte, North Carolina
  - Barrett Cancer, Cincinnati, Ohio
  - CORTPA, Dallas, Texas
  - Urology of Virginia-Sentara Medical Group, Norfolk, Virginia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Amin A, Dudek AZ, Logan TF, Lance RS, Holzbeierlein JM, Knox JJ, Master VA, Pal SK, Miller WH Jr, Karsh LI, Tcherepanova IY, DeBenedette MA, Williams WL, Plessinger DC, Nicolette CA, Figlin RA. Survival with AGS-003, an autologous dendritic cell-based immunotherapy, in combination with sunitinib in unfavorable risk patients with advanced renal cell carcinoma (RCC): Phase 2 study results. J Immunother Cancer. 2015 Apr 21;3:14. doi: 10.1186/s40425-015-0055-3. eCollection 2015. PMID 25901286
- See also: Argos Therapeutics Website — http://www.argostherapeutics.com
- See also: Kidney Cancer Association — http://www.nkca.org